CLINICAL TRIAL: NCT03983382
Title: A Safety and Feasibility Study of Limited Cardiac Monitoring During Non-anthracycline Trastuzumab-based Therapy in Patients With HER2-positive Breast Cancer
Brief Title: A Study of Limited Heart Monitoring During Non-anthracycline Trastuzumab-based Therapy in Breast Cancer Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 19-045
Record Dates: First submitted 2019-06-07; First posted 2019-06-12 (Actual); Results first posted 2024-10-28 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
Keywords: non-anthracycline trastuzumab; trastuzumab; Memorial Sloan Kettering Cancer Center; 19-045
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HER2-Positive Breast Cancer
  Interventions: Diagnostic Test: Left Ventricular Ejection Fraction

INTERVENTIONS:
Diagnostic Test: Left Ventricular Ejection Fraction — LVEF assessment at baseline, 6 months, and 12 months
  Other Names: LVEF

SUMMARY:
The purpose of this study is to test whether patients with breast cancer who are being treated with non-anthracycline trastuzumab therapy can safely be monitored for heart related side effects less often than usual.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years
* Newly diagnosed histologically confirmed primary invasive breast carcinoma (Stage I-IV)
* Pathologically confirmed HER2-positive breast cancer
* Planned to receive trastuzumab-based therapy for a minimum of 12 months, or started trastuzumab-based therapy within the last weeks with a planned duration of at least 12 months.
* Normal LV systolic function (EF greater than or equal to the institutional lower limit of normal)
* William and able to comply with the requirements of the protocol

Exclusion Criteria:

* Planned to receive an anthracycline-based regimen
* Prior history of treatment with anthracycline chemotherapy
* History of cardiovascular including cardiomyopathy, heart failure, or any other clinically significant cardiovascular disease (as determined by the investigator)
* Uncontrolled hypertension, defined as systolic blood pressure >/= 160 mmHg and/or diastolic blood pressure >/= 90 mmHg (as determined by the investigator)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A member of the patient's treatment team, the protocol investigator, or research team at MSK will identify potential research participants. The preliminary screen of eligibility will be confirmation of the diagnosis of HER2-positive breast cancer. A member of the treatment team will discuss the study and the possibility of enrollment in the study with potential subjects that meet this eligibility criterion. The study will be conducted at the Evelyn H. Lauder Breast Center of MSK as well as at the regional MSK network sites. Recruitment at both main and regional network sites will ensure the enrollment of diverse populations of different ages, races, and ethnic groups onto the study. Patients will then be consented to the study.
  In most cases, the initial contact with the prospective subject will be conducted either by the treatment team, investigator or the research staff working in consultation with the treatment team.
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2026-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Yu, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Hartford Healthcare Cancer Institute @ Hartford Hospital (Data collection only), Hartford, Connecticut
  - Memorial Sloan Kettering Cancer Center @ BaskingRidge (Consent and follow-up only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent and Follow up), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent and follow-up only), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Commack (Consent and Follow up), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent and Follow-up), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Consent and Follow-up), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
• Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Derived] Yu AF, Dang CT, Jorgensen J, Moskowitz CS, DeFusco P, Oligino E, Oeffinger KC, Liu JE, Steingart RM. Rationale and design of a cardiac safety study for reduced cardiotoxicity surveillance during HER2-targeted therapy. Cardiooncology. 2023 Mar 9;9(1):13. doi: 10.1186/s40959-023-00163-4. PMID 36895062
- See also: Memorial Sloan Kettering Cancer Center — http://mskcc.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HER2-Positive Breast Cancer
Started | 190
Completed | 172
Not Completed | 18
Not completed — Death | 1
Not completed — Lost to Follow-up | 3
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 10
Not completed — Change in cancer treatment | 2

BASELINE CHARACTERISTICS:
Arm/Group | HER2-Positive Breast Cancer
Number analyzed (Participants) | 190
Age, Continuous [Mean (Full Range); unit: years] | 52 [24 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 190
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18
  Not Hispanic or Latino | 158
  Unknown or Not Reported | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 24
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 139
  More than one race | 0
  Unknown or Not Reported | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 190

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Cardiac Adverse Events, Defined by a Compositive of Clinical Heart Failure (NYHA Class III or IV) or Cardiac Death.
Time Frame: 12 months from baseline
Measure: Number; unit: Cardiac AEs
Arm/Group | HER2-Positive Breast Cancer
Number analyzed (Participants) | 190
Cardiac AEs | 0

ADVERSE EVENTS:
Time Frame: 1 years
Arm/Group | HER2-Positive Breast Cancer
All-Cause Mortality (participants affected / at risk) | 1/190
Serious Adverse Events (participants affected / at risk) | 1/190
Other Adverse Events (participants affected / at risk) | 8/190
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HER2-Positive Breast Cancer (N=190)
Death NOS (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HER2-Positive Breast Cancer (N=190)
Left ventricular- systolic dysfunction (Cardiac disorders) | 1
Cardiac Disorders- Other specify (Cardiac disorders) | 3
Edema: Limb (General disorders) | 2
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Ventricular arrhythmia-Ventricular tachycardia (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-07): https://cdn.clinicaltrials.gov/large-docs/82/NCT03983382/Prot_SAP_000.pdf